CLINICAL TRIAL: NCT00807092
Title: Comparison of the Efficacy on Glycaemic Control and Safety Profile of Biphasic Insulin Aspart 30 and Biphasic Human Insulin 30 Both in Combination With Metformin in Insulin-naïve Subjects With Type 2 Diabetes Mellitus Inadequately Controlled on Oral Antidiabetic Drugs (OADs) Therapy
Brief Title: Comparing the Efficacy and Safety of Biphasic Insulin Aspart 30 and Biphasic Human Insulin 30 on Blood Sugar Control in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-3681
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2011-04-11 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; biphasic human insulin 30; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIAsp 30 (Experimental): BIAsp 30 (biphasic insulin aspart 30) administered subcutaneously (under the skin) twice daily (before breakfast and dinner) + metformin. Initial total daily dose of 0.3 U or IU/kg body weight followed by individual dose adjustment for BIAsp 30 was performed over the first 4 weeks (titration period) to achieve the pre-meal blood glucose target of 4.4-6.1 mmol/l. The achieved dose was maintained for the last 2 weeks of treatment unless hypoglycaemia occurred.
  Interventions: Drug: biphasic insulin aspart 30; Drug: metformin
- BHI 30 (Experimental): BHI 30 (biphasic human insulin 30) administered subcutaneously (under the skin) twice daily (30 minutes before breakfast and dinner) + metformin. Initial total daily dose of 0.3 U or IU/kg body weight followed by individual dose adjustment for BHI 30 was performed over the first 4 weeks (titration period) to achieve the pre-meal blood glucose target of 4.4-6.1 mmol/l. The achieved dose was maintained for the last 2 weeks of treatment unless hypoglycaemia occurred.
  Interventions: Drug: biphasic human insulin 30; Drug: metformin

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — The initial doses for BIAsp 30 twice-daily regimen will be recommended to start at a total daily dose of 0.3 U/kg body weight and to be equally divided (1/2:1/2) between pre-breakfast and pre-dinner
  Arms: BIAsp 30
Drug: biphasic human insulin 30 — The initial doses for BHI 30 twice-daily regimen will be recommended to start at a total daily dose of 0.3 IU/kg body weight and to be divided in the ratio of 2/3:1/3 between pre-breakfast and pre-dinner
  Arms: BHI 30
Drug: metformin — Metformin dose must remain the same as that used prior to the trial.

SUMMARY:
This trial is conducted in Asia. The aim of this clinical trial is to investigate the blood sugar lowering effect and the safety profile of biphasic insulin aspart 30 compared to biphasic human insulin 30, both in combination with metformin in Chinese insulin-naive subjects with type 2 diabetes when failing on oral antidiabetic drug (OAD) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosed for at least 6 months
* Insulin-naive (less than or equal to 1 week of daily use of insulin therapy)
* Treatment with metformin as monotherapy or in combination therapy with other OAD(s) for at least 3 months prior to this trial
* Currently on metformin greater than or equal to 1000 mg/day for at least 2 weeks
* Currently at least one of other OAD(s) reaching at least one-half of the recommended maximum dose for at least 2 weeks
* Glycosylated haemoglobin (HbA1c) between 7.5-11.0%
* Body Mass Index (BMI) between 18.5 - 35.0 kg/m^2
* Be able and willing to perform continuous glucose monitoring system (CGMS ) and self-monitored blood glucose (SMBG)

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products
* Any contraindication of metformin
* Receipt of investigational drug within the last 3 months prior to this trial
* Any history of chronic insulin therapy (more than 1 week of daily use)
* Systemically treated with thiazolidinediones (TZDs) for more than one month within 6 months prior to this trial
* Pregnancy, nursing mother, or unwillingness to use adequate contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Beijing, Beijing Municipality, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 10 sites across China
Pre-assignment Details: All eligible subjects had their baseline blood glucose profiles monitored by continuous glucose monitoring system (CGMS) for 72 hours. Following CGMS uninstall and discontinuation of all previous oral anti-diabetic drug (OAD) treatment, subjects were randomised to one of two treatment groups.
Period: Overall Study
Arm/Group | BIAsp 30 | BHI 30
Started | 72 | 73
Exposed to Drug | 71 (Subject was randomised, but not exposed to any trial drug) | 73
Completed | 71 | 69
Not Completed | 1 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — CGMS data collection failed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIAsp 30 | BHI 30 | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (9) | 54.4 (10.4) | 55.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 39 | 72
  Male | 38 | 34 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 71 | 73 | 144
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 66.28 (12) | 65.49 (11.4) | 65.88 (11.7)
Height at screening [Mean (Standard Deviation); unit: m] | 1.634 (0.09) | 1.623 (0.09) | 1.628 (0.09)
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 24.68 (3) | 24.74 (3) | 24.71 (3)
Duration of diagnosed diabetes [Mean (Standard Deviation); unit: years] | 7.74 (5.5) | 7 (5.2) | 7.36 (5.3)
HbA1c at screening [Mean (Standard Deviation); unit: percentage of total haemoglobin] | 9.19 (1.05) | 9.08 (1.08) | 9.13 (1.06)
Metformin monotherapy or combination therapy at randomisation [Number; unit: participants] — OAD treatment at randomisation
  participants
    Metformin Monotherapy | 20 | 18 | 38
    Metformin Combination Therapy | 51 | 55 | 106

OUTCOME MEASURES:

1. Primary Outcome: Change in IAUC (Incremental Area Under the Curve) for Postprandial Glucose (0-4 Hours) Over 3 Main Meals
Description: The blood glucose profiles were monitored by CGMS (Continuous Glucose Monitoring System) for 72 hours at baseline (week 0) and end of treatment (week 6). IAUC was calculated using the trapezoidal method. The arithmetic mean of IAUC (3 meal-specific incremental areas) of day 1 and day 2 was used as the value of IAUC for each CGMS period
Time Frame: Week 0, week 6
Population: The full analysis set using LOCF (Last Observation Carried Forward) consists of all randomised subjects who had been exposed to at least one dose of the trial products.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 30 | BHI 30
Number analyzed (Participants) | 67 | 63
mmol/L | -1.99 (0.49) | -1.977 (0.517)
Statistical Analysis 1: Comparison: BIAsp 30 vs BHI 30; The null hypothesis (H0) was: H0: Change in mean IAUC(0-4hours) of BIAsp 30 after 6 weeks of treatment-Change in mean IAUC(0-4hours) of BHI 30 after 6 weeks of treatment greater than or equal to 0 mol*h/L against the alternative hypothesis(H1): H1: Change in mean IAUC (0-4hours) of BIAsp 30 after 6 weeks of treatment-Change in mean IAUC(0-4hours) of BHI 30 after 6 weeks of treatment less than 0 mol*h/L; Test type: Superiority or Other; ANCOVA — A statistical significant threshold p less than 0.025; Treatment and strata as factors; baseline (visit 2) value of mean IAUC(0-4hours) as covariate; Mean Difference (Net) = -0.013, 95% CI [-1.332 to 1.306], Standard Error of Mean 0.666 — BIAsp 30 - BHI 30

2. Secondary Outcome: Change in Mean IAUC for Postprandial Glucose (0-4 Hours) After Each Meal (Breakfast, Lunch, Dinner) Assessed by CGMS
Description: The blood glucose profiles were monitored by CGMS for 72 hours at baseline (week 0) and end of treatment (week 6). IAUC (0-4 hours) after each meal at 6 weeks and change in IAUC (0-4 hours) from baseline (week 0) after each meal were to be assessed. The arithmetic mean of day 1 and day 2 for each meal-specific incremental area (breakfast, lunch, dinner) was calculated.
Time Frame: Week 0, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 30 | BHI 30
Number analyzed (Participants) | 71 | 73
mmol/L
  Breakfast, N=68, 64 | -3.094 (0.725) | -4.272 (0.765)
  Lunch, N=69, 66 | 1.651 (0.897) | 1.969 (0.93)
  Dinner, N=69, 65 | -4.775 (0.539) | -4.026 (0.566)
Statistical Analysis 1: Comparison: BIAsp 30 vs BHI 30; Null hypothesis and alternative hypothesis for breakfast: The null hypothesis (H0) was: H0: Change in mean IAUC(0-4h) of BIAsp 30 for breakfast after 6 weeks of treatment-Change in mean IAUC(0-4h) of BHI 30 for breakfast after 6 weeks of treatment =0 mol*h/L against the alternative hypothesis(H1): H1: Change in mean IAUC (0-4h) of BIAsp 30 for breakfast after 6 weeks of treatment-Change in mean IAUC(0-4h) of BHI 30 for breakfast after 6 weeks of treatment≠0 mol*h/L; Test type: Superiority or Other; p = 0.2412, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; corresponding baseline (week 0) value of mean IAUC(0-4h) as covariate (breakfast/lunch/dinner); Mean Difference (Net) = 1.178, 95% CI [-0.802 to 3.157], Standard Error of Mean 1 — Breakfast
Statistical Analysis 2: Comparison: BIAsp 30 vs BHI 30; Null hypothesis and alternative hypothesis for lunch: The null hypothesis (H0) was: H0: Change in mean IAUC(0-4h) of BIAsp 30 for lunch after 6 weeks of treatment-Change in mean IAUC(0-4h) of BHI 30 for lunch after 6 weeks of treatment =0 mol*h/L against the alternative hypothesis(H1): H1: Change in mean IAUC (0-4h) of BIAsp 30 for lunch after 6 weeks of treatment-Change in mean IAUC(0-4h) of BHI 30 for lunch after 6 weeks of treatment≠0 mol*h/L; Test type: Superiority or Other; p = 0.794, ANCOVA — A statistical significant threshold p<0.05; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.318, 95% CI [-2.724 to 2.087], Standard Error of Mean 1.216 — Lunch
Statistical Analysis 3: Comparison: BIAsp 30 vs BHI 30; Null hypothesis and alternative hypothesis for dinner: The null hypothesis (H0) was: H0: Change in mean IAUC(0-4h) of BIAsp 30 for dinner after 6 weeks of treatment-Change in mean IAUC(0-4h) of BHI 30 for dinner after 6 weeks of treatment =0 mol*h/L against the alternative hypothesis(H1): H1: Change in mean IAUC (0-4h) of BIAsp 30 for dinner after 6 weeks of treatment-Change in mean IAUC(0-4h) of BHI 30 for dinner after 6 weeks of treatment≠0 mol*h/L; Test type: Superiority or Other; p = 0.3093, ANCOVA — A statistical significant threshold p<0.05; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -0.749, 95% CI [-2.2 to 0.703] — Dinner

3. Secondary Outcome: Mean FBG (Fasting Blood Glucose) Assessed by CGMS
Description: The blood glucose profiles were monitored by CGMS for 72 hours at end of treatment (week 6). Mean FBG assessed by CGMS at 6 weeks. FBG was read on the CGMS glucose curves at 06:00 each morning over the 72 hours. The arithmetic mean of day 1 and day 2 was used as the value of mean FBG for each CGMS period.
Time Frame: Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 30 | BHI 30
Number analyzed (Participants) | 69 | 66
mmol/L | 6.861 (0.193) | 6.414 (0.2)
Statistical Analysis 1: Comparison: BIAsp 30 vs BHI 30; The null hypothesis (H0) was: H0: Change in mean FBG of BIAsp 30 after 6 weeks of treatment-Change in mean FBG of BHI 30 after 6 weeks of treatment =0 mmol/L against the alternative hypothesis(H1): H1: Change in mean FBG of BIAsp 30 after 6 weeks of treatment-Change in mean FBG of BHI 30 after 6 weeks of treatment≠0 mmol/L; Test type: Superiority or Other; p = 0.0891, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of mean FBG as covariate; Mean Difference (Net) = 0.448, 95% CI [-0.069 to 0.964], Standard Error of Mean 0.261

4. Secondary Outcome: Change in Mean FBG Assessed by CGMS
Description: The blood glucose profiles were monitored by CGMS for 72 hours at baseline (week 0) and at end of treatment (week 6). Change in mean FBG from baseline (week 0) was assessed. FBG was read on the CGMS glucose curves at 06:00 each morning over the 72 hours. The arithmetic mean of day 1 and day 2 was used as the value of mean FBG for each CGMS period.
Time Frame: Week 0, week 6
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 30 | BHI 30
Number analyzed (Participants) | 69 | 66
mmol/L | -2.114 (0.193) | -2.561 (0.2)

5. Secondary Outcome: Change in FPG (Fasting Plasma Glucose)
Description: FPG was analysed by local laboratories at baseline (week 0) and end of treatment (week 6). Change in FPG at end of treatment (week 6) from baseline (week 0) was to be assessed.
Time Frame: Week 0, Week 6
Population: The full analysis set using LOCF (Last Observation Carried Forward) (if a measurement on the withdrawal visit was available) consists of all randomised subjects who had been exposed to at least one dose of the trial products.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 30 | BHI 30
Number analyzed (Participants) | 70 | 68
mmol/L | -2.961 (0.185) | -3.456 (0.188)
Statistical Analysis 1: Comparison: BIAsp 30 vs BHI 30; The null hypothesis (H0) was: H0: Change in FPG of BIAsp 30 after 6 weeks of treatment-Change in FPG of BHI 30 after 6 weeks of treatment =0 mmol/L against the alternative hypothesis(H1): H1: Change in FPG of BIAsp 30 after 6 weeks of treatment-Change in FPG of BHI 30 after 6 weeks of treatment≠0 mmol/L; Test type: Superiority or Other; p = 0.0472, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of mean FBG as covariate; Mean Difference (Net) = 0.495, 95% CI [0.0060 to 0.984], Standard Error of Mean 0.247

6. Secondary Outcome: Change in 8-point SMBG (Self-monitored Blood Glucose) Profiles
Description: Subjects were asked to perform 8-point SMBG profiles using the provided blood glucose meter on one day within 72 hours CGMS monitoring period at week 0 and week 6. Change in blood glucose level at end of treatment (week 6) from baseline (week 0) at each time point was to be assessed respectively. Blood glucose levels were measured at the following 8 time points: Before each meal (breakfast, lunch and dinner), 120 minutes after the start of each meal, at bedtime and at 3 am in the morning.
Time Frame: Week 0, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 30 | BHI 30
Number analyzed (Participants) | 71 | 73
mmol/L
  Before Breakfast, N=71, 68 | -2.27 (0.2) | -2.38 (0.2)
  2 hours after Breakfast, N=69, 69 | -3.99 (0.41) | -5.22 (0.41)
  Before Lunch, N=71, 68 | -3.46 (0.3) | -3.73 (0.31)
  2 hours after Lunch, N=70, 69 | -2.24 (0.38) | -2.41 (0.39)
  Before dinner, N=70, 69 | -2.59 (0.36) | -2.32 (0.37)
  2 hours after Dinner, N=70, 69 | -4.57 (0.36) | -4.1 (0.36)
  Bedtime, N=71, 68 | -3.84 (0.3) | -4.03 (0.31)
  3AM, N=68, 66 | -2.62 (0.21) | -3.39 (0.22)
  Average, N=71, 69 | -3.16 (0.18) | -3.43 (0.19)
Statistical Analysis 1: Comparison: BIAsp 30 vs BHI 30; For each endpoint of SMBG :The null hypothesis (H0) was: H0: Change in BG of BIAsp 30 after 6 weeks of treatment-Change in BG of BHI 30 after 6 weeks of treatment =0 mmol/L against the alternative hypothesis(H1): H1: Change in BG of BIAsp 30 after 6 weeks of treatment-Change in BG of BHI 30 after 6 weeks of treatment≠0 mmol/L; Test type: Superiority or Other; p = 0.676, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 2) value of BG as covariate; Mean Difference (Net) = 0.11, 95% CI [-0.41 to 0.63] — Before breakfast
Statistical Analysis 2: Comparison: BIAsp 30 vs BHI 30; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.026, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of BG as covariate; Mean Difference (Net) = 1.23, 95% CI [0.15 to 2.31] — 2 hours after breakfast
Statistical Analysis 3: Comparison: BIAsp 30 vs BHI 30; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.5, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of BG as covariate; Mean Difference (Net) = 0.27, 95% CI [-0.53 to 1.08] — Before lunch
Statistical Analysis 4: Comparison: BIAsp 30 vs BHI 30; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.747, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of BG as covariate; Mean Difference (Net) = 0.17, 95% CI [-0.86 to 1.19] — 2 hours after lunch
Statistical Analysis 5: Comparison: BIAsp 30 vs BHI 30; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.581, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of BG as covariate; Mean Difference (Net) = -0.27, 95% CI [-1.23 to 0.69] — Before dinner
Statistical Analysis 6: Comparison: BIAsp 30 vs BHI 30; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.326, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of BG as covariate; Mean Difference (Net) = -0.47, 95% CI [-1.42 to 0.48] — 2 hours after dinner
Statistical Analysis 7: Comparison: BIAsp 30 vs BHI 30; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.643, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of BG as covariate; Mean Difference (Net) = 0.19, 95% CI [-0.61 to 0.99] — Bedtime
Statistical Analysis 8: Comparison: BIAsp 30 vs BHI 30; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0080, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of BG as covariate; Mean Difference (Net) = 0.77, 95% CI [0.21 to 1.33] — 3 AM
Statistical Analysis 9: Comparison: BIAsp 30 vs BHI 30; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.274, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of BG as covariate; Mean Difference (Net) = 0.27, 95% CI [-0.22 to 0.75] — Average

7. Secondary Outcome: Change in Prandial Blood Glucose Increment
Description: Subjects were asked to perform 8-point SMBG profiles using the provided blood glucose meter on one day within 72 hours CGMS monitoring period at week 0 and week 6 respectively. Prandial increment was the difference between the blood glucose (BG) value measured 120 minutes after meal and the BG value measured before meal.
Time Frame: Week 0, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 30 | BHI 30
Number analyzed (Participants) | 71 | 73
mmol/L
  Breakfast, N=69, 68 | -1.82 (0.39) | -2.82 (0.4)
  Lunch, N=70, 68 | 1.32 (0.44) | 1.27 (0.45)
  Dinner, N=69, 69 | -1.91 (0.42) | -1.85 (0.42)
  Average, N=70, 68 | -0.81 (0.21) | -1.1 (0.22)
Statistical Analysis 1: Comparison: BIAsp 30 vs BHI 30; For each endpoint of Prandial Blood Glucose Increment :The null hypothesis (H0) was: H0: Change in prandial BG increment of BIAsp 30 after 6 weeks of treatment-Change in prandial BG increment of BHI 30 after 6 weeks of treatment =0 mmol/L against the alternative hypothesis(H1): H1: Change in prandial BG increment of BIAsp 30 after 6 weeks of treatment-Change in prandial BG increment of BHI 30 after 6 weeks of treatment≠0 mmol/L; Test type: Superiority or Other; p = 0.062, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of prandial BG increment as covariate; Mean Difference (Net) = 0.99, 95% CI [-0.05 to 2.04] — Breakfast
Statistical Analysis 2: Comparison: BIAsp 30 vs BHI 30; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.933, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of prandial BG increment as covariate; Mean Difference (Net) = 0.05, 95% CI [-1.12 to 1.22] — Lunch
Statistical Analysis 3: Comparison: BIAsp 30 vs BHI 30; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.922, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of prandial BG increment as covariate; Mean Difference (Net) = -0.05, 95% CI [-1.16 to 1.05] — Dinner
Statistical Analysis 4: Comparison: BIAsp 30 vs BHI 30; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.313, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of prandial BG increment as covariate; Mean Difference (Net) = 0.29, 95% CI [-0.28 to 0.85] — Average

8. Secondary Outcome: Change in MAGE (Mean Amplitude of Glycaemic Excursions) Assessed by CGMS
Description: MAGE is a parameter to monitor the intraday blood glucose excursions. It was calculated using CGMS data and as the arithmetic mean of glycaemic excursion with the criterion that both segments (ascending and descending parts) of the glycaemic excursion exceed of the value of one standard deviation of respective 24-hour blood glucose value. The direction of calculation (peak-to-nadir or nadir-to-peak) was established by the direction of the first excursion. The arithmetic mean of the glycaemic excursion of day 1 and day 2 was the value of MAGE for each CGMS
Time Frame: Week 0, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | BIAsp 30 | BHI 30
Number analyzed (Participants) | 69 | 69
mmol/L | -0.499 (0.273) | -0.686 (0.284)
Statistical Analysis 1: Comparison: BIAsp 30 vs BHI 30; The full analysis set using LOCF (Last Observation Carried Forward) consists of all randomised subjects who had been exposed to at least one dose of the trial products; Test type: Superiority or Other; p = 0.6149, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (visit 2) value of mean MAGE as covariate; Mean Difference (Net) = 0.187, 95% CI [-0.547 to 0.921], Standard Error of Mean 0.371

9. Secondary Outcome: Change in GA (Glycated Albumin)
Description: Glycated Albumin is used as a general glycaemic control parameter. Analysed by laboratory. GA was measured at baseline (week 0) and end of treatment (week 6). Change in GA at end of treatment (week 6) from baseline (week 0) was assessed.
Time Frame: Week -2, week 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage point change
Arm/Group | BIAsp 30 | BHI 30
Number analyzed (Participants) | 70 | 68
percentage point change | -6.147 (0.428) | -6.474 (0.438)
Statistical Analysis 1: Comparison: BIAsp 30 vs BHI 30; The null hypothesis (H0) was: H0: Change in GA of BIAsp 30 after 6 weeks of treatment-Change in GA of BHI 30 after 6 weeks of treatment =0 % against the alternative hypothesis(H1): H1: Change in GA of BIAsp 30 after 6 weeks of treatment-Change in GA of BHI 30 after 6 weeks of treatment≠0 %; Test type: Superiority or Other; p = 0.5706, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of GA as covariate; Mean Difference (Net) = 0.328, 95% CI [-0.813 to 1.468], Standard Error of Mean 0.577

10. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Time Frame: Week -2, week 6
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage point change
Arm/Group | BIAsp 30 | BHI 30
Number analyzed (Participants) | 71 | 68
percentage point change | -1.647 (0.083) | -1.667 (0.086)
Statistical Analysis 1: Comparison: BIAsp 30 vs BHI 30; The null hypothesis (H0) was: H0: Change in HbA1c of BIAsp 30 after 6 weeks of treatment-Change in HbA1c of BHI 30 after 6 weeks of treatment =0 % against the alternative hypothesis(H1): H1: Change in HbA1c of BIAsp 30 after 6 weeks of treatment-Change in HbA1c of BHI 30 after 6 weeks of treatment≠0%; Test type: Superiority or Other; p = 0.8598, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of HbA1c as covariate; Mean Difference (Net) = 0.02, 95% CI [-0.243 to 0.243], Standard Error of Mean 0.113

11. Secondary Outcome: Duration of Hypoglycaemic Events Based on CGMS
Description: The CGMS device recorded blood glucose levels every 10 seconds then stored a smoothed average over 5 minutes. The range of blood glucose detection was 2.2-22 mmol/l. Hypoglycaemia was defined as blood glucose readings below 3.5 mmol/l or below 2.5 mmol/l, respectively. The duration of the hypoglycaemic episodes was quantified by accumulating the total time the CGMS profiles stays below the defined threshold (i.e. below 3.5 mmol/l or below 2.5 mmol/l, respectively).
Time Frame: 72-hour monitoring period at Week 0 and Week 6
Population: Safety analysis set consists of all randomised subjects who were exposed to at least one dose of trial product(s).
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | BIAsp 30 | BHI 30
Number analyzed (Participants) | 71 | 73
Hours
  Blood glucose < 3.5 mmol/L, N=70, 68 | 0.304 (0.094) | 0.358 (0.097)
  Blood glucose < 2.5 mmol/L, N=70, 68 | 0.048 (0.028) | 0.06 (0.029)
Statistical Analysis 1: Comparison: BIAsp 30 vs BHI 30; The null hypothesis (H0) was: H0: Duration of Hypoglycaemic Events Based on CGMS of BIAsp 30 after 6 weeks of treatment-Duration of Hypoglycaemic Events Based on CGMS of BHI 30 after 6 weeks of treatment =0 hours against the alternative hypothesis(H1): H1: Duration of Hypoglycaemic Events Based on CGMS of BIAsp 30 after 6 weeks of treatment-Duration of Hypoglycaemic Events Based on CGMS of BHI 30 after 6 weeks of treatment≠0 hours; Test type: Superiority or Other; p = 0.671, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of duration of hypoglycaemic events as covariate; Mean Difference (Net) = -0.054, 95% CI [-0.307 to 0.198], Standard Error of Mean 0.128 — Blood glucose below 3.5 mmol/l
Statistical Analysis 2: Comparison: BIAsp 30 vs BHI 30; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.7544, ANCOVA — A statistical significant threshold p<0.05; Treatment and strata as factors; baseline (week 0) value of duration of hypoglycaemic events as covariate; Mean Difference (Net) = -0.012, 95% CI [-0.088 to 0.064], Standard Error of Mean 0.038 — Blood glucose below 2.5 mmol/l

12. Secondary Outcome: Hypoglycaemia Based on Self-reported Episodes
Description: Total number of hypoglycaemic episodes occurring in the trial after baseline (week 0) until the end of treatment (week 6). Hypoglycaemic episodes are classified as major, minor or symptoms only: Major if the subject was unable to treat her/himself; minor if subject was able to treat her/himself and self monitored blood glucose (SMBG) was below 2.8 mmol/L; symptoms only if subject was able to treat her/himself and with no blood glucose measurement or SMBG higher than or equal to 2.8 mmol/L.
Time Frame: Weeks 0-6
Population: Safety analysis set consists of all randomised subjects who were exposed to at least one dose of trial product(s).
Measure: Number; unit: episodes
Arm/Group | BIAsp 30 | BHI 30
Number analyzed (Participants) | 71 | 73
episodes
  All | 63 | 55
  Major | 3 | 3
  Minor | 9 | 10
  Symptoms only | 51 | 42

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time span of 6 weeks (starting from the start of treatment to the end of treatment plus one day)
Description: The safety analysis set contains all randomised subjects exposed to at least one dose of trial drug(s).
Arm/Group | BIAsp 30 | BHI 30
Serious Adverse Events (participants affected / at risk) | 1/71 | 3/73
Other Adverse Events (participants affected / at risk) | 0/71 | 0/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIAsp 30 (N=71) | BHI 30 (N=73)
Loose body in joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 2 (2)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to not release data until specified milestones. This includes the right to not release interim results of clinical trials. At the end of the trial, manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.